CLINICAL TRIAL: NCT05173896
Title: Improving Cerebral Blood Flow and Cognition in Patients with Cerebral Small Vessel Disease. the ETLAS-2 Trial
Acronym: ETLAS2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christina Kruuse (Other)
Collaborators: Danish Research Centre for Magnetic Resonance (Other); Bispebjerg Hospital (Other); Rigshospitalet, Denmark (Other); University of Copenhagen (Other); The Novo Nordic Foundation (Other); Nordsjaellands Hospital (Other)
Responsible Party: Sponsor-Investigator, Christina Kruuse, MD, Ph.D., DMSc, Professor in Neurology, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-20031301; 2020-002329-27 (EudraCT Number)
Record Dates: First submitted 2021-11-16; First posted 2021-12-30 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Small Vessel Diseases; Stroke, Ischemic
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Ischemic Stroke | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tadalafil (Experimental): Oral tadalafil (20 mg) capsules once daily for three months.
  Interventions: Drug: Tadalafil 20 MG
- Placebo (Placebo Comparator): Oral placebo capsules once daily for three months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil 20 MG — Daily dose of oral over-encapsulated tadalafil tablets (20 mg) for three months.
  Arms: Tadalafil
Drug: Placebo — Daily dose of oral over-encapsulated placebo tablets for three months.
  Arms: Placebo

SUMMARY:
In a randomized controlled trial the feasibility and effect of three months treatment with daily tadalafil, on cerebral blood flow/reactivity and cognition, is investigated in patients with cerebral small vessel disease.

DETAILED DESCRIPTION:
Cerebral small vessel disease is a progressive brain and blood vessel disease for which there currently is no effective treatment. The disease associates with 25 % of all stroke and 30 % of all dementia cases and imposes a major and increasing health burden worldwide. In this trial the investigator suggest a new promising solution to this problem.

Patients with cerebral small vessel disease, who experience stroke or vascular dementia, may show reduced brain perfusion or altered neurovascular reactivity. The investigator has previously shown that a single dose of tadalafil (20 mg), shortly increased blood supply to the brain in patients with cerebral small vessel disease. This holds promise for new effective treatment targets. The investigator test if patients find three months daily intake of tadalafil (20 mg) feasible, and if it alters cerebral perfusion, neurovascular reactivity, and cognition, including memory and planning ability. The trial will help identify new treatment targets to reduce the number of patients with stroke, stroke sequelae, and vascular dementia.

This trial is divided into one main study and three sub studies:

* Main study
* Dynamical MRI sub study
* Cognitive sub study
* Biomarker sub study

ELIGIBILITY:
Inclusion Criteria:

1. MRI/computed tomography (CT) evidence of small vessel occlusion stroke(s)/lacunar stroke(s) (involving ≤2 cm in the acute phase and ≤1.5cm in the late phase) and/or confluent deep white matter hyperintensities (≥ grade 2 on Fazekas's scale).
2. Clinical evidence of cerebral small vessel disease can be: a) small vessel occlusion stroke (lacunar stroke) syndrome with symptoms lasting > 24 hours, occurring < 5 years ago; OR b) transient ischemic attack (TIA) with symptoms lasting < 24 hours AND with MR-DWI imaging performed acutely showing small vessel occlusion stroke, occurring < 5 years ago; OR c) TIA with symptoms lasting < 24 hours AND no acute MRI-DWI lesion but MRI/CT evidence of CSVD with old small vessel occlusion stroke(s) (involving ≤1.5cm) and/or confluent deep white matter hyperintensities (≥ grade 2 on Fazekas's scale).
3. Age ≥ 50 years.

Exclusion Criteria:

1. Known diagnosis of dementia, medically treated dementia, or under investigation for dementia
2. Pregnancy or nursing
3. Women of childbearing age not taking contraception
4. Known cortical infarction (> 1.5 cm maximum diameter)
5. Known carotid artery stenosis ≥ 50 % with Doppler ultrasound, CT angiography, or MRI angiography diagnosed within the last five years
6. Known carotid or vertebral dissection as a cause of stroke
7. Stroke after carotid or heart surgery
8. Known hypercoagulable disease
9. Systolic BP < 90 and/or diastolic BP < 50
10. Known severe renal impairment (eGFR < 30ml/min)
11. Known severe hepatic impairment (Child-Pugh > B)
12. History of non-arthritic anterior ischemic optic neuropathy
13. Concomitant use of PDE5 inhibitors e.g. sildenafil, tadalafil, and vardenafil during trial period
14. Patients receiving nicorandil and nitrates e.g. isosorbide mononitrate, isosorbide dinitrate, glyceryl trinitrate
15. History of acute myocardial infarction in the last three months before trial intervention
16. Body weight > 130kg
17. Known cardiac failure (NYHA ≥ II)
18. Known persistent or paroxysmal atrial fibrillation/flutter
19. History of "sick sinus syndrome" or other supraventricular cardiac conduction conditions such as sinoatrial or atrioventricular block (2nd of 3rd degree)
20. Other known cardiogenic cause of stroke
21. Contraindication to CO2 challenge, eg severe respiratory disease
22. MRI not tolerated or contraindicated
23. Known monogenic causes of stroke i.e. CADASIL
24. Unable to provide informed consent
25. The participant does not wish to be informed about results from the MRI

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of treatment defined as proportion of participants achieving full target dose of tadalafil/placebo. | From baseline to three months.
  Number of participants achieving full target dose of tadalafil/placebo by end of three months trial period. Outcome will be assessed by a structured questionnaire with tablet count.

SECONDARY OUTCOMES:
MRI - Cerebral Blood Flow | From baseline to three months.
  Change in cerebral blood flow measured with arterial spin labeling (ASL) during a sensory hand stimulus.
MRI - Neurovascular reactivity and perfusion | From baseline to three months.
  Change in neurovascular reactivity, coupling, and cerebral blood flow/perfusion measured with BOLD/ASL during a visual stimulation with and without a carbon dioxide vascular challenge.
MRI - Neurovascular reactivity | From baseline to three months.
  Change in neurovascular reactivity measured with blood-oxygen-level dependent (BOLD) during a sensory hand stimulus.
MRI - Blood Brain Barrier | From baseline to three months.
  Change in blood brain barrier measured with diffusion-prepared (DP)-ASL MRI.
MRI - STRIVE criteria | From baseline to three months.
  Relative changes (%) in STRIVE assessment, including new strokes, white matter hyperintensity, cerebral microbleeds, enlarged perivascular space, atrophy, and lacunes.
Montreal Cognitive Assessment | From baseline to three months.
  Change in Montreal Cognitive Assessment (MoCA) score. Score range 0-30. Higher scores mean a better outcome.
Symbol Digit Modalities Test | From baseline to three months.
  Change in Symbol Digit Modalities Test (SDMT) score. Score range 0-110. Higher scores mean a better outcome.
Dementia Assessment by Rapid Test | From baseline to three months.
  Change in Dementia Assessment by Rapid Test - DART score. Score range 0-50. Higher scores mean a better outcome.
Trail Making Test A | From baseline to three months.
  Change in time to perform Trail Making Test A. Quicker time means a better outcome.
Trail Making Test B | From baseline to three months.
  Change in time to perform Trail Making Test B. Quicker time means a better outcome.
Digit Span Forward | From baseline to three months.
  Change Digit Span Forward test score. Score range 0-16. Higher scores mean a better outcome.
Digit Span Backward | From baseline to three months.
  Change Digit Span Backward test score. Score range 0-16. Higher scores mean a better outcome.
Digit Span Arrangement | From baseline to three months.
  Change Digit Span Arrangement test score. Score range 0-16. Higher scores mean a better outcome.
WAIS Letter Number Sequence | From baseline to three months.
  Change Letter Number sequence test score. Score range 0-30. Higher scores mean a better outcome.
Word mobilising test - F, S, A, and animals | From baseline to three months.
  Change word mobilising test score. Higher scores mean a better outcome.
Cambridge Neuropsychological Test Automated Battery - Spatial Working Memory | From baseline to three months.
  Change in spatial working memory score.
Cambridge Neuropsychological Test Automated Battery - Motor Screening | From baseline to three months.
  Change in motor screening score.
Cambridge Neuropsychological Test Automated Battery - Rapid Visual Information processing | From baseline to three months.
  Change in rapid visual information processing score.
Cambridge Neuropsychological Test Automated Battery - Paired Associates Learning Task | From baseline to three months.
  Change in paired associates learning task score.
Cambridge Neuropsychological Test Automated Battery - One-Touch Stockings of Cambridge | From baseline to three months.
  Change in One-Touch Stockings of Cambridge score.
Cambridge Neuropsychological Test Automated Battery - Reaction Time | From baseline to three months.
  Change in reaction time score.
Short Informant Questionnaire on Cognitive Decline in the Elderly - IQCODE | From baseline to three months.
  Change in short IQCODE score. Score range 1-5. A score of 3 means that the subject is rated on average as 'no change'.
Becks Depression Inventory - BDD | From baseline to three months.
  Change in BDD score. Score range 0-63. Higher score means increased risk of depression.
Fatigue Severity Scale - FSS | From baseline to three months.
  Change in FSS score. Score range 0-7. Higher score means increased fatigue severity.
WHO-5 Well-Beeing Index | From baseline to three months.
  Change in WHO-5 score. Score range 0-100. Higher score means better quality of life.
Vascular- and inflammatory biomarkers: vascular cell adhesion molecule (VCAM-1) | From baseline to three months.
  Changes in vascular cell adhesion molecule (VCAM-1) (unit pg/ml).
Vascular- and inflammatory biomarkers: intercellular adhesion molecule-1 (ICAM-1) | From baseline to three months.
  Changes in intercellular adhesion molecule-1 (ICAM-1) (unit pg/ml).
Vascular- and inflammatory biomarkers: interleukin-6 (IL-6) | From baseline to three months.
  Changes in interleukin-6 (IL-6) (unit pg/ml).
Vascular- and inflammatory biomarkers: tumour necrosis factor alpha (TNF-α) | From baseline to three months.
  Changes in tumour necrosis factor alpha (TNF-α) (unit pg/ml).
Vascular- and inflammatory biomarkers: interleukin 1beta (IL-1β) | From baseline to three months.
  Changes in interleukin 1beta (IL-1β) (unit pg/ml).
Vascular- and inflammatory biomarkers: E-selectin | From baseline to three months.
  Changes in E-selectin (unit pg/ml).
Vascular- and inflammatory biomarkers: vascular endothelial growth factor (VEGF) | From baseline to three months.
  Changes in vascular endothelial growth factor (VEGF) (unit pg/ml).
Vascular- and inflammatory biomarkers: specific micro RNA | From baseline to three months.
  Changes in specific micro RNA associated to vascular disease.
Death, ischemic and hemorrhagic event, and dementia | From baseline to five years.
  Difference in composite measure of death, any ischemic event, hemorrhagic event or dementia per patient registry after three and five years respectively from end of trial.
Blood pressure | From baseline to three months.
  Change in both systolic and diastolic blood pressure (unit mmHg).
Heart rate | From baseline to three months.
  Change in heart rate (unit beats per minute).
Adverse events | From baseline to three months.
  Difference in adverse events between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Kruuse, MD, Prof, Principal Investigator — Herlev Gentofte Hospital, Department of Neurology
Locations (2):
- Denmark (2):
  - Department of Neurology, Herlev Gentofte Hospital, Herlev
  - Danish Research Centre for Magnetic Resonance, Hvidovre

IPD SHARING:
Plan to Share IPD: Yes
IPD can be accessed upon reasonable request and after evaluation from the investigator.

REFERENCES:
- [Derived] Olmestig J, Mortensen KN, Thomas MB, Fagerlund B, Robbins TW, Naveed N, Nordling MM, Christensen H, Iversen HK, Poulsen MB, Siebner HR, Kruuse C. Cognitive outcomes after tadalafil treatment in patients with cerebral small vessel disease: ETLAS-2 sub-study. Cereb Circ Cogn Behav. 2025 Nov 11;9:100520. doi: 10.1016/j.cccb.2025.100520. eCollection 2025. PMID 41332889
- [Derived] Olmestig J, Mortensen KN, Thomas MB, Fagerlund B, Naveed N, Nordling MM, Nielsen MKK, Rasmussen BS, Christensen H, Iversen HK, Poulsen MB, Siebner HR, Kruuse C. Tadalafil Treatment in Patients With Cerebral Small Vessel Disease: The ETLAS-2 Randomized Clinical Trial. Stroke. 2025 Oct;56(10):2846-2857. doi: 10.1161/STROKEAHA.125.051602. Epub 2025 Jul 28. PMID 40718899
- [Derived] Olmestig J, Mortensen KN, Fagerlund B, Naveed N, Nordling MM, Christensen H, Iversen HK, Poulsen MB, Siebner HR, Kruuse C. Cerebral blood flow and cognition after 3 months tadalafil treatment in small vessel disease (ETLAS-2): study protocol for a randomized controlled trial. Trials. 2024 Aug 29;25(1):570. doi: 10.1186/s13063-024-08402-4. PMID 39210472